CLINICAL TRIAL: NCT02572388
Title: Safety and Immunogenicity of a Protein Particle Malaria Vaccine Candidate, R21, Administered With and Without Matrix-M1 in Healthy UK Volunteers
Brief Title: A Study to Assess the Safety and Immunogenicity of the Malaria Vaccine, R21, Administered With and Without Matrix-M1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC053
Record Dates: First submitted 2015-10-01; First posted 2015-10-08 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-01

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — R21 monoclonal antibody; Matrix-M

ARMS (4):
- Group 1 (Active Comparator): 10µg of R21 mixed with 50µg of Matrix-M on days 0, 28, and 56.
  Interventions: Biological: R21; Biological: Matrix-M1
- Group 2 (Active Comparator): 50µg of R21 on days 0, 28, and 56.
  Interventions: Biological: R21
- Group 3 (Active Comparator): 50µg of R21 mixed with 50µg of Matrix-M on days 0, 28, and 56.
  Interventions: Biological: R21; Biological: Matrix-M1
- Group 4 (Active Comparator): 2µg of R21 mixed with 50µg of Matrix-M
  Interventions: Biological: R21; Biological: Matrix-M1

INTERVENTIONS:
Biological: R21
Biological: Matrix-M1
  Arms: Group 1; Group 3; Group 4

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered one or two experimental malaria vaccines. The vaccine R21 will either be administered alone or in combination with the adjuvant vaccine Matrix-M1.

All vaccinations will be administered intramuscularly. Each volunteer will receive three vaccinations in total.

There are three different vaccine schedules:

Group 1 will receive 10µg of R21 mixed with 50µg of Matrix-M1 on days 0, 28, and 56.

Group 2 will receive 50µg of R21 on days 0, 28, and 56. .

Group 3 will receive 50µg of R21 mixed with 50µg of Matrix-M1 on days 0, 28, and 56.

The study will assess the safety of the vaccines, and the immune responses to the vaccinations. Immune responses are measured by tests on blood samples.

Healthy adult volunteers will be recruited in Oxford and London, England.

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
* Any history of anaphylaxis in relation to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* History of clinical malaria (any species)
* Travel to a malaria endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, Oxfordshire
  - NIHR Wellcome Trust Clinical Research Facility, Hammersmith Hospital, London

REFERENCES:
- [Derived] Venkatraman N, Tiono AB, Bowyer G, Bellamy DG, Stockdale LK, Powlson J, Collins KA, Coulibaly S, Datoo MS, Silman D, Ouedraogo A, Nebie I, Imoukhuede EB, Brod F, Folegatti P, Dickinson-Craig E, Jamieson S, Bougouma EC, Wright D, Diarra A, Bliss CM, Morter R, Glenn G, Fries LF, Reimer JM, Lovgren-Bengtsson K, Baker M, Poulton I, Moyle S, Berrie E, Green N, Mukhopadhyay E, Viebig NK, Angus B, Lawrie A, Roberts R, Gilbert SC, Lewis DJM, Sirima SB, Ewer KJ, Hill AVS. Evaluation of a novel malaria anti-sporozoite vaccine candidate, R21 in Matrix-M adjuvant, in the UK and Burkina Faso: two phase 1, first-in-human trials. Lancet Microbe. 2025 Mar;6(3):100868. doi: 10.1016/S2666-5247(24)00084-3. Epub 2025 Jan 10. PMID 39805302

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 10µg of R21 mixed with 50µg of Matrix-M on days 0, 28, and 56.
  R21
  Matrix-M1
- Group 2: 50µg of R21 on days 0, 28, and 56.
  R21
- Group 3: 50µg of R21 mixed with 50µg of Matrix-M on days 0, 28, and 56.
  R21
  Matrix-M1
- Group 4: 2µg of R21 mixed with 50µg of Matrix-M
  R21
  Matrix-M1
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 11 | 4 | 10 | 6
Completed | 10 | 3 | 8 | 4
Not Completed | 1 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 11 | 4 | 10 | 6 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 4 | 10 | 6 | 31
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 5 | 2 | 16
  Male | 4 | 2 | 5 | 4 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 4 | 10 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Administration of R21 With and Without the Adjuvant Matrix-M1 Assessed by the Occurrence of Solicited Local and Systemic Adverse Events.
Description: Occurrence of solicited local and systemic adverse events (i.e: pain, redness, swelling and pruritus at injection site and temperature, feverishness, myalgia, arthralgia, malaise, headache and nausea).
Time Frame: Assessment of solicited AEs in the first 7 days post vaccination.
Measure: Number; unit: Number of Adverse Events per group
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 11 | 4 | 10 | 6
Number of Adverse Events per group | 103 | 21 | 94 | 21

2. Primary Outcome: Safety and Tolerability of R21 With and Without the Adjuvant Matrix-M1 Assessed by the Occurrence of Unsolicited Adverse Events.
Description: Occurrence of unsolicited local and systemic adverse events.
Time Frame: Unsolicited AEs to be assessed up to 28 days post vaccination.
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 11 | 4 | 10 | 6
participants | 11 | 4 | 10 | 6

3. Primary Outcome: Safety and Tolerability of R21 With and Without the Adjuvant Matrix-M1 Assessed by the Occurrence of Serious Adverse Events.
Description: Occurrence of serious adverse events collected from enrolment until the end of the follow-up period.
Time Frame: 6 months
Population: There is no SAEs in groups 2 and 3
Measure: Number; unit: Number of Serious AEs
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 11 | 4 | 10 | 6
Number of Serious AEs | 1 | 0 | 0 | 1

4. Primary Outcome: Safety and Tolerability of R21 With and Without the Adjuvant Matrix-M1 Assessed by the Occurrence of Laboratory Adverse Events.
Description: Occurrence of laboratory adverse events defined as clinically significant changes from baseline. Haematology (Full Blood Count) and Biochemistry (Kidney and Liver Function Tests) will be assessed.
Time Frame: At Day 0 (baseline), day 7 and day 28 post vaccination
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 11 | 4 | 10 | 6
participants | 11 | 4 | 10 | 6

ADVERSE EVENTS:
Time Frame: Solicited adverse events will be recorded daily for 7 days post-vaccination Unsolicited AEs of all severities will be recorded from receipt of vaccination through 28 days post-vaccination. After study Day 28, only SAEs or new chronic medical conditions that require ongoing medical management will be recorded through to the last study visit.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/4 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/4 | 0/10 | 1/6
Other Adverse Events (participants affected / at risk) | 10/11 | 3/4 | 9/10 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=11) | Group 2 (N=4) | Group 3 (N=10) | Group 4 (N=6)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=11) | Group 2 (N=4) | Group 3 (N=10) | Group 4 (N=6)
Pain (General disorders) | 10 (10) | 3 (3) | 9 (9) | 3 (3) — Vaccination 1
Headache (General disorders) | 4 (4) | 1 (1) | 3 (3) | 0 (0) — Vaccination 1
Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Vaccination 1
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Vaccination 1
Itch (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Vaccination 1
Warmth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) — Vaccination 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0) — Vaccination 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Vaccination 1
Feverishness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) — Vaccination 1
Fatigue (General disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (1) — Vaccination 1
Nausea (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — Vaccination 1
Malaise (General disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) — Vaccination 1
Pain (General disorders) | 10 (10) | 3 (3) | 7 (7) | 2 (2) — Vaccination 2
Redness (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) — Vaccination 2
Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Vaccination 2
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — Vaccination 2
Warmth (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) — Vaccination 2
Fever (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Vaccination 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) — Vaccination 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Vaccination 2
Feverishness (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) — Vaccination 2
Headache (General disorders) | 4 (4) | 1 (1) | 4 (4) | 2 (2) — Vaccination 2
Fatigue (General disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1) — Vaccination 2
Nausea (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) — Vaccination 2
Malaise (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) — Vaccination 2
Pain (General disorders) | 8 (8) | 1 (1) | 6 (6) | 2 (2) — Vaccination 3
Redness (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 2 (2) | 2 (2) — Vaccination 3
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Vaccination 3
Itch (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Vaccination 3
Warmth (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) — Vaccination 3
Feverishness (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Vaccination 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 3 (3) | 0 (0) — Vaccination 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Vaccination 3
Headache (General disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (1) — Vaccination 3
Fatigue (General disorders) | 4 (4) | 0 (0) | 5 (5) | 0 (0) — Vaccination 3
Nausea (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Vaccination 3
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Vaccination 3
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Vaccination 1
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) — Vaccination 2
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Vaccination 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT02572388/Prot_SAP_000.pdf